CLINICAL TRIAL: NCT05647421
Title: A Comparative Study of Visual Outcome of Two Extended Depth of Focus Intraocular Lenses After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Badawy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-43-2022
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Visual To Compare the Visual Outcome Between AcrySof™ IQ Vivity™ and TECNIS Synergy™ Intraocular Lens (Model ZFR00V )

STUDY DESIGN:
Intervention Model Description: AcrySof™ IQ Vivity™ and TECNIS Synergy™ Intraocular Lens (Model ZFR00V )
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The AcrySof™ IQ Vivity™ intraocular lens group (Active Comparator): The AcrySof™ IQ Vivity™ will be implanted in 20 eyes of 10 patients (group 1)
  Interventions: Device: IOL implantation
- TECNIS Synergy™ Intraocular Lens (Model ZFR00V ) group (Active Comparator): The TECNIS Synergy™ Intraocular Lens (Model ZFR00V ) will be implanted in 20 eyes of 10 patients
  Interventions: Device: IOL implantation

INTERVENTIONS:
Device: IOL implantation — after phacoemulsification of the cataract , implantation of Acrysof IQVIVITY IOL .
Device: IOL implantation — after phacoemulsification of the cataract , implantation of TECNIS Synergy™ Intraocular Lens (Model ZFR00V )

SUMMARY:
The investigators aim to compare the visual performance of the most recently introduced extended depth of focus intraocular lenses ; AcrySofTM IQ VivityTM and TECNIS SynergyTM ( an extended depth of focus IOL ) regarding the range of vision (using defocus curve ) , contrast sensitivity( through the modulation transfer function curves ) and their effect on ocular aberrations as the ivestigators believe that proper study of these aspects could influence the investigators choice and guidance to the cataract patient about the most suitable presbyopia correcting IOL .

DETAILED DESCRIPTION:
Presbyopia-correcting IOLs can be divided into 4 broad categories: Enhanced monofocal IOLs , Mutifocal IOLs (including diffractive or refractive designs) , extended depth-of-focus (EDOF) IOLs, and accommodative IOLs .

Standard multifocal lenses ( e.g : FineVision® (Physiol, Liège, Belgium) are diffractive IOLs which split incident light into two or more points of focus, but these lenses are limited by the optical aberrations and the presence of secondary out-of-focus image and photic phenomena .

The new Tecnis® EyhanceIOL (model ICB00, Johnson & Johnson Vision, Santa Ana, CA, USA) is a refractive modified monofocal lens with better intermediate visual acuity than standard monofocal IOLs and eliminates the dysphotopsia that is common with the standard multifocal IOLs and compensates for the spherical aberration of the cornea due to its high order aspheric profile .

The EDOF IOL, or extended range of vision IOL, incorporates a new technology which createsa single-elongated focal point to enhance the depth-of-focus, contrary to monofocal IOLs (in which light is focused on one single point) or MF IOLs (having 2 or 3 discrete points). This elongated focus is introduced to eliminate the overlapping of near and far images caused by traditional MF IOLs, thus eliminating the halo effect .However , EDOF IOLs are thought to be inferior to standard trifocal IOls regarding near vision.

AcrySof™ IQ Vivity™ Extended Vision Intraocular Lens (Alcon, Fort Worth, Texas,USA ) was approved by the Food and Drug Administration in February 2020 and it is considered the most recently introduced non-diffractive EDOF IOL . TECNIS Synergy™ Intraocular Lens (Model ZFR00V) (Johnson & Johnson Vision,SantaAna, CA, USA) is a continuous depth of focus intraocular lens and was approved by food and drug administration in April 2021 . it combines both elements of standard multifocal and extended depth of focus with preservation of high contrast sensitivity .

The investigators aim to compare the visual performance of the most recently introduced extended depth of focus intraocular lengths ; AcrySof™ IQ Vivity™ and TECNIS Synergy™ ( an extended depth of focus IOL ) regarding the range of vision (using defocus curve ) , contrast sensitivity( through the modulation transfer function curves ) and their effect on ocular aberrations as the investigators believe that proper study of these aspects could influence the ophthalmologists' choice and guidance to the cataract patient about the most suitable presbyopia correcting IOL .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery.
* Preoperative corneal astigmatism equal to or less than 0.75 D

Exclusion Criteria:

* Other ocular comorbidities which may affect the outcome of our research such as glaucoma, corneal opacities , chronic or recurrent anterior uveitis, diabetic retinopathy , age -related macular degeneration.
* Previous ocular surgeries

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Range of vision of the different IOLs represented by the defocus curve | within 1 month after surgery
  monocular defocus curve will be obtained by using the best corrected distance refraction and measuring the visual acuity Between +1.50 D and- 2.50 D in 0.5-D defocus steps, except in the region from +0.50 D through* 0.50 D, which would be done in -0.25D steps. Letters will be randomly presented to avoid memorization.

SECONDARY OUTCOMES:
Contrast sensitivity (which will be objectively assessed through modulation transfer function ) - Photic phenomena (which will be objectively expressed through the ocular aberration ). | within 1 month after the surgery
  Modulation transfer function under mesopic eye condition and total ocular aberrations will be assessed using ITrace aberrometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanclerz P, Toto F, Grzybowski A, Alio JL. Extended Depth-of-Field Intraocular Lenses: An Update. Asia Pac J Ophthalmol (Phila). 2020 May-Jun;9(3):194-202. doi: 10.1097/APO.0000000000000296. PMID 32511121
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Auffarth GU, Gerl M, Tsai L, Janakiraman DP, Jackson B, Alarcon A, Dick HB; Quantum Study Group. Clinical evaluation of a new monofocal IOL with enhanced intermediate function in patients with cataract. J Cataract Refract Surg. 2021 Feb 1;47(2):184-191. doi: 10.1097/j.jcrs.0000000000000399. PMID 32932369
- [Background] Kohnen T, Herzog M, Hemkeppler E, Schonbrunn S, De Lorenzo N, Petermann K, Bohm M. Visual Performance of a Quadrifocal (Trifocal) Intraocular Lens Following Removal of the Crystalline Lens. Am J Ophthalmol. 2017 Dec;184:52-62. doi: 10.1016/j.ajo.2017.09.016. Epub 2017 Sep 18. PMID 28923587
- [Background] Carballo-Alvarez J, Vazquez-Molini JM, Sanz-Fernandez JC, Garcia-Bella J, Polo V, Garcia-Feijoo J, Martinez-de-la-Casa JM. Visual outcomes after bilateral trifocal diffractive intraocular lens implantation. BMC Ophthalmol. 2015 Mar 14;15:26. doi: 10.1186/s12886-015-0012-4. PMID 25884715